CLINICAL TRIAL: NCT02023684
Title: Routine Irrigation With Ropivacaine vs. Lidocaine vs. Saline of Surgical Bed in Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Principal Investigator, Hagar Mizrahi, Doctor, The Baruch Padeh Medical Center, Poriya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 10-2013.CTIL
Record Dates: First submitted 2013-11-08; First posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-11

CONDITIONS: Overweight and Obesity
Keywords: Sleeve Gastrectomy; Lidocaine; ropivacaine
MeSH Terms: conditions — Overweight; Obesity | interventions — Sodium Chloride; Lidocaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control (Placebo Comparator): Irrigation will be carried out with saline
  Interventions: Drug: control saline
- Lidocaine (Active Comparator): Irrigation will be carried out with Lidocaine
  Interventions: Drug: Lidocaine
- Ropivacaine (Active Comparator): Irrigation will be carried out with Ropivacaine
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: control saline — Surgical bed irrigation with saline 40ml
  Other Names: saline
  Arms: control
Drug: Lidocaine — surgical bed Irrigation Lidocaine 0.5%, 40ml
  Arms: Lidocaine
Drug: Ropivacaine — surgical bed Irrigation Ropivacaine 0.2%, 40ml
  Arms: Ropivacaine

SUMMARY:
The aim of this study is to evaluate the effect of ropivacaine and lidocaine irrigation at the surgical bed on postoperative pain relief and breathing parameters in laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
As in any other surgery, postoperative pain control after bariatric procedure should provide comfort and early mobilisation as well as enable adequate respiratory effort.

Early ambulation is thought to reduce the risk of pressure ulcers, deep vein thrombosis and respiratory complications. In contrast, early inadequate postoperative pain management can lead to hypoxemia, hypercarbia and atelectasis. However, the use of opioids for pain control is limited in bariatric surgery due to sedative effect which might worsen obstructive sleep apnoea (OSA), a common comorbidity amongst morbidly obese patients and opioid-sparing techniques might help avoid respiratory complications.

Methods of regional analgesic are limited and might be challenging in the obese patient and although techniques such continuous epidural analgesia is possible it is not the common practise. The use of patient-controlled i.v. analgesia of opioids is limited owed to increased risk for hypoxemia and other practises such as routine local anaesthetic port site wound infiltration and systemic non-steroidal drugs are warranted.

The benefit of intra-peritoneal irrigation with local anaesthetic for abdominal pain relief after laparoscopic procedures was established in few studies. The aim of this study is to evaluate the effect its' effect on postoperative pain relief and breathing parameters in laparoscopic sleeve gastrectomy.By pain score

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to sleeve gastrectomy

Exclusion Criteria:

* Second bariatric procedure Patients younger than 18 years Patients who have drug allergy to Lidocaine or Ropivacain Patients who suffer a cardiac arrhythmia Pregnant patients Mentally challenged patients Patients who refuse to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The aim of the study is to evaluate the effect of local irrigation with ropivacaine vs. Lidocaine vs. Saline of surgical bed in sleeve gastrectomy on post operative pain | 1 year
  measuring the score of pain using visual analog score for pain during the post-operative timemeasuring the number of times pain-control durg were given during the post-operate time

CONTACTS AND LOCATIONS:
Overall Officials: Hagar Mizrahi, M.D. MSc, Principal Investigator — The BARUCH PADEH Medical Center, Poriya, ISRAEL
Locations (1):
- General Surgery Ward, Poria – Neve Oved, The Lower Galilee, Israel